CLINICAL TRIAL: NCT05017558
Title: Operational Evaluation of the Introduction of "Point Of Care" (POC) to Optimise Post-natal Prophylaxis of HIV-exposed Newborns According to the Risk of Maternal to Child Transmission (MTCT) Assessed by Measuring Maternal Viral Load at Delivery in Conakry, Guinea
Brief Title: Evaluation of Measurement of Maternal Viral Load at Delivery to Optimise Post-natal Prophylaxis of HIV-exposed Newborns
Acronym: IPOP
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Responsible Party: Sponsor
Other Study IDs: ANRS12412 IPOP
Record Dates: First submitted 2021-07-19; First posted 2021-08-24 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Mother to Child HIV Transmission
Keywords: prevention of mother to child HIV transmission; HIV early diagnosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- intervention: Measurement of viral load in HIV-1 infected mothers at delivery by POC to optimise post-natal prophylaxis and neonatal diagnosis of children according to the estimated risk of MTCT (high risk:VL at delivery ≥ 1000 copies/mL, low risk: VL at delivery < 1000 copies/mL) in Conakry, Guinea.
  Interventions: Diagnostic Test: point of care

INTERVENTIONS:
Diagnostic Test: point of care — HIV-1 infected women will benefit from a viral load measurement by POC (Cepheid GenXpert HIV-1 viral load) at the time of delivery.
  Newborns will benefit :
  1. Antiretroviral preventive treatment differentiated according to their risk of infection in accordance with national recommendations:
     * High risk (maternal VL ≥1000 cp/ml): AZT/NVP for 12 weeks.
     * Low risk (maternal VL <1000 cp/ml): NVP for 6 weeks.
  2. virological screening for HIV by qualitative POC (Cepheid GenXpert HIV-1 qual) from birth (for high-risk newborns) at 6 weeks, at 9 months and at any time in the event of clinical manifestations suggestive of HIV infection.
  3. In the event of a positive HIV test, the child will initiate immediately AZT/3TC/LPV/r
  4. support from volunteers to improve retention in care, promotion of exclusive breastfeeding and family nutritional support

SUMMARY:
The main objective is to evaluate the operationality of introducing the measurement of viral load in HIV-1 infected mothers at delivery by POC to optimise post-natal prophylaxis and neonatal diagnosis of children according to the estimated risk of MTCT (high risk: HIV viral load (VL) at delivery ≥ 1000 copies/mL, low risk: VL at delivery < 1000 copies/mL) in Conakry, Guinea.

DETAILED DESCRIPTION:
Intervention:

All women screened for HIV-1 infection in the delivery room, whether or not the infection was previously known, whether or not they are treated, will be eligible to participate in this study and will be offered inclusion in the study.

The women will benefit from a viral load measurement by POC (Cepheid GenXpert HIV-1 viral load) at the time of delivery.

Newborns will benefit :

1. the provision of antiretroviral (ARV) preventive treatment differentiated according to their risk of infection in accordance with national recommendations:

   * High risk (maternal VL ≥1000 cp/ml): zidovudine (AZT)/ nevirapine (NVP) for 12 weeks.
   * Low risk (maternal VL <1000 cp/ml): NVP for 6 weeks.
2. early and regular virological screening for HIV by qualitative POC (Cepheid GenXpert HIV-1 qual) from birth (for high-risk newborns) at 6 weeks, at 9 months and at any time in the event of clinical manifestations suggestive of HIV infection.
3. In the event of a positive HIV test, the child will initiate immediate antiretroviral treatment combining zidovudine (AZT)/ lamivudine (3TC)/ Lopinavir-retonivir (LPV/r) and a confirmatory test will be done by POC (Cepheid GenXpert HIV-1 viral load) according to World Health Organisation (WHO) and national recommendations.
4. support from the project team and peers, volunteers from the association Fédération Espoir Guinée (FEG), to improve retention in care and compliance of mother and child, promotion of exclusive breastfeeding for 6 months and family nutritional support, Cotrimoxazole (CTX) prophylaxis and the Expanded Programme on Immunization will be provided by the national programme.

ELIGIBILITY:
Inclusion Criteria:

* For mother:
* Mother/child couple whose mother is HIV-1 infected, whether or not the infection is known and treated at delivery
* Mother of full age 18 years or older
* Mother agreeing to be contacted by telephone to ensure that appointments are respected.
* Mother has signed the informed consent form to participate in the study (and agrees to be followed, along with her child, at the centre for the duration of the study).

For children:

* Live newborn baby
* Free, informed and written consent must be signed by the holder(s) of parental authority and the investigator for the child's participation in this research (at the latest on the day of birth and before any intervention carried out on the newborn in the trial).

Exclusion Criteria:

For mother:

* Mother infected with HIV-2
* Not included due to monitoring difficulties:

  * Anticipated absence(s) that could hinder participation in research (travel abroad, relocation, travel);
  * Insufficient motivation to be followed for 9 months in the centre.
  * No mobile phone or refusal to be called by investigators if necessary.
* Mother and/or children already participating in another biomedical study

For children:

* Not included for reasons of caution (child with severe congenital malformation or clinical symptomatology suggesting opportunistic infection).
* The child has a known allergy to the drug given as part of HIV prophylaxis in Guinea or to its components.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Measurement of viral load in HIV-1 infected mothers at delivery by POC to optimise post-natal prophylaxis and neonatal diagnosis of children according to the estimated risk of MTCT (high risk:VL at delivery ≥ 1000 copies/mL, low risk: VL at delivery < 1000 copies/mL) in Conakry, Guinea.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-03 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Evaluate the operationally of introducing the measurement of viral load in HIV-1 infected mothers at delivery by POC | Day 0 to day 2
  Proportion of newborns having received antiretroviral prophylaxis within 48 hours after delivery adapted to the "real" risk of MTCT, defined by measuring the maternal viral load by POC at delivery.

SECONDARY OUTCOMES:
To evaluate the intrinsic diagnostic performance of viral load measurement by POC Xpert HIV-1 in comparison with the evaluation of the level of risk by maternal interrogation alone. | Day 0 to day 2
  Sensitivity and specificity of the risk level assessment by the interrogation data in comparison with viral load measurement as a reference method.
  Defining the level of risk through interrogation :
  * High risk: newborn of an HIV-infected mother who is not treated with antiretroviral (ARV) within 4 weeks before delivery and/or who discovers HIV infection at delivery;
  * Low risk: newborn of HIV-infected mother treated with ARV since ≥ 4 weeks before delivery).
  Defining the level of risk by measuring HIV viral load:
  * High risk: VL>1000 cp/mL
  * Low risk: VL≤ 1000 cp/mL
To assess the proportion of women who received Xpert HIV-1 viral load test at delivery. | Day 0 to day 2
  Proportion of women who received Xpert HIV-1 viral load test at delivery.
To assess the turn around time of Xpert HIV-1viral load | Day 0 to day 2
  Total time (day) from sampling to result of Xpert HIV-1 viral load test performed at delivery
To measure the satisfaction of health care staff and mothers with the use of the POC test to monitor viral load in mothers. | Day 0 to day 2
  Measure, through a questionnaire, the satisfaction of health workers and mothers with the use of the POC test to monitor viral load in mothers. for mothers the questionnaires will be analyzed on a scale of 0 to 25 , with a score of 25 corresponding to maximum satisfaction. For health workers the questionnaires will be analyzed on a scale of 8 to 32, with a score of 32 corresponding to maximum satisfaction.
To assess the proportion of children who received Xpert HIV-1 qual test | Day 0 to week 9
  Proportion of children who received Xpert HIV-1 qual test at birth for children at high risk, and at week 6 and week 9 for all children
To assess the turn around time of Xpert HIV-1 qual test | Day 0 to week 9
  Total time (day) from sampling to result of Xpert HIV-1 qual test at birth for children at high risk, and at week 6 and week 9 for all children
To measure the satisfaction of health care workers and mothers with the use of the POC test for early infant diagnosis. | Day 0 to week 9
  Measure, through a questionnaire, the satisfaction of health workers and mothers with the use of the POC test to monitor viral load in mothers. for mothers the questionnaires will be analyzed on a scale of 0 to 25 , with a score of 25 corresponding to maximum satisfaction. For health workers the questionnaires will be analyzed on a scale of 8 to 32, with a score of 32 corresponding to maximum satisfaction.
To collect feedback from health professionals and mothers on the use of POC in the clinic. | Day 0 to week 9
  collect feedback from health professionals and mothers on the use of POC in the clinic, during individual interview at the end of the study.
To assess the proportion of women ready to start or continue ARV treatment ("ARV readiness") during the study, comparing the proportion of women lost to follow-up from day 0 to month 9. | Day 0 to month 9
  Measure the proportion of women ready to start or continue ART ("ARV readiness") during the study using a questionnaire, comparing the proportion of women lost to follow-up from day 0 to month 9.
  The questionnaires will be analyzed on a scale of 5 to 25, with a score of 25 corresponding to the highest readiness to initiate the treatment.
To determine whether the stigma of the women included in the study affects the proportion lost to follow-up during the study. | Week 6 to month 9
  Determine using a questionnaire administered at 6 weeks whether stigma of the women included in the study affects the proportion lost to follow-up during the study, by comparing data from month 3 and month 9 to week 6. The questionnaires will be analyzed on a scale of 0 to 13, with a score of 13 corresponding to maximum stigmatisation level.
To assess the proportion of untreated women initiating ARV treatment | Day 0 to day 2
  Proportion of untreated women initiating ARV treatment at day 0 at the time of delivery
To assess the proportion of women lost to follow-up | Day 0 to month 9
  Proportion of HIV-1 infected women lost to follow-up between day 0 and month 9
To assess the proportion of HIV-1 infected women with virological success | Month 6
  Proportion of mothers whose HIV viral load is <1000 cp/mL and <50 cp/mL at month 6
To assess the proportion of children lost to follow-up | Day 0 to month 9
  Proportion of children lost to follow-up from day 0 to month 9
To assess the proportion of HIV-1 infected children initiating ARV treatment | Day 0 to month 9
  Proportion of children with a diagnosis of HIV infection made between day 0 and month 9, initiating ARV treatment.
To assess the turn around time from from sample collection to ARV treatment initiation in HIV-1 infected children | Day 0 to month 9
  Delay between sample collection and initiation of ARV treatment in the case of diagnosis of HIV infection in children from day 0 to month 9.
To assess the rate of mother-to-child transmission of HIV | Day 0 to month 9
  Proportion of HIV-infected children between day 0 and month 9 among children followed from day 0 to month 9 whose HIV status is known.
To assess the proportion of women practicing exclusive breastfeeding. | Day 0 to month 6
  Proportion of women reporting exclusive breastfeeding up to month 6.
To measure, in women with a VL<1000 cp/mL at delivery who do not report taking ARV, the proportion of those with ARV detectable in the plasma and the nature of those ARV detected. | Day 0 to day 2
  Proportion of women with VL <1000 and reporting not taking ARV, having ARV detectable in plasma and the nature of these ARV
To measure, in women with a VL>1000 cp/mL at delivery and reporting taking ARV, the proportion of those with ARV detectable in the plasma and the nature of these ARV detected. | Day 0 to day 2
  Proportion of women with VL ≥1000 at delivery and reporting taking ARV, having plasma-detectable ARVs and the nature of these ARV
To measure the proportion of women reporting taking ARV before childbirth and having a detectable VL at delivery, the proportion of viruses with ARV resistance mutations. | Day 0 to day 2
  Proportion of women with detectable VL (≥ 50 cp/mL) at delivery whose virus has ARV resistance mutations and the nature of these mutations.
To measure the proportion of HIV-infected children with ARV resistance mutations. | Day 0 to month 9
  Proportion of children infected with HIV whose virus has ARV resistance mutations and the nature of these mutations.
Assess patient adherence to ARV treatment on the basis of adherence questionnaires from day 0 to months 9 | Day 0 to 9 month 9
  Proportion of women on ARV treatment reporting less than 2 uptake left per week on day 0 (for women on pre-delivery treatment only), month 3, month 6 and months 9.
Assess patient adherence to ARV treatment on the basis of ARV dosage at day 0 (only for mothers treated before delivery) and at month 6. | Day 0 to month 6
  Proportion of patients on treatment in whom ARV were detected in plasma at effective residual concentration at day 0 (for women on treatment before delivery only), and at month 6.
Socio-anthropological survey: Assessment of feelings about the study among mothers, fathers, psychosocial counsellors and health professionals. | 9 months
  Evaluation, by means of individual interviews at the end of the study, of the feelings of mothers, fathers, psychosocial counsellors and health professionals about the study.

IPD SHARING:
Plan to Share IPD: Undecided